CLINICAL TRIAL: NCT05492084
Title: Personalized Risk of Rapidly Progressive Atherosclerosis
Acronym: RPA
Status: Completed | Type: Observational
Sponsor: Novosibirsk State Medical University (Other)
Collaborators: Novosibirsk State University (Other)
Responsible Party: Principal Investigator, Natalya G. Lozhkina, professor of the Novosibirsk State Medical University, Novosibirsk State Medical University
Other Study IDs: L-001
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Atherosclerosis, Coronary
Keywords: rapidly progressive atherosclerosis; personalized risk
MeSH Terms: conditions — Coronary Artery Disease | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — frozen blood clot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- active group: The first - active group (100 people) included patients who had type 1 myocardial infarction (MI) (54 people) within 2 years prior to the study or the diagnosis of CAD was established according to selective coronary angiography: the presence lumen stenosis of at least two coronary arteries by 50 % or more (46 people) and an additional two (or more) cardiovascular events from the following: MI or unstable angina, emergency arterial stenting, stroke, peripheral arterial thrombosis, critical ischemia, and lower limb amputation. The combination of two or more of these cardiovascular events that occurred within two years indicated the rapid progression of atherosclerosis in these patients.
  Interventions: Other: without Intervention
- comparison group: The second (comparison group) included 102 patients with confirmed coronary heart disease in a similar way (55 people had only 1 type 1 MI in the past and 45 had coronary artery disease confirmed by selective coronary angiography, respectively), in whom two years before inclusion in the study there were no cardiovascular events from the above, which indicated the spontaneous course of atherosclerosis.
  Interventions: Other: without Intervention

INTERVENTIONS:
Other: without Intervention — without Intervention

SUMMARY:
Вackground. Progressive atherosclerosis is accompanied by unfavorable clinical outcomes, study and understanding of this process, creation of risk assessment method is necessary for individualization of approaches to treatment and prevention of this condition.

Purpose of the study. Creation of a mathematical model to assess the risk of accelerated atherosclerosis development, using methods of factor and correlation analysis.

Patient Characteristics and Study Methods. A retrospective cohort study included 202 patients with coronary heart disease. Group 1 included patients who had had myocardial infarction or unstable angina, emergency arterial stenting, stroke, peripheral artery thrombosis, critical ischemia, and lower extremity amputation within 2 years before study inclusion. Patients in the comparison group did not have these events. The influence of each of the studied parameters on the probability of fast progressing atherosclerosis was determined by factor and correlation analysis. The prospective part of the study will include follow-up of patients from both groups for 12 months. Annual "endpoints": fatal outcome, unscheduled coronary revascularization, nonfatal myocardial infarction and stroke, hospitalization due to unstable angina pectoris, stent thrombosis, stenting/plasty of lower limb arteries.

DETAILED DESCRIPTION:
Study design: open continuous retrospective and prospective study by parallel group method.

Three control points were defined in the dissertation work: the first point was retrospective, 2 years before the study; the second was the day of inclusion in the study; and the third was 12 months after inclusion.

The retrospective point covered 2 years from the date of patient inclusion in the study (period from January 2019 to January 2021) with determination of a large spectrum of parameters of clinical, instrumental, laboratory nature potentially influencing the appearance and progression of atherosclerosis (according to the literature analysis). The mentioned examinations were performed and evaluated at two points: the first one - at the time of the first preceding coronary event during the two-year retrospective period, the second one - at the time of the patient's inclusion in the present study. 202 patients were divided into two groups.

Study Methods. At the moment of inclusion (1 point) in the study all patients underwent general clinical examination with assessment of complaints and clinical status, laboratory examination with general and biochemical blood tests, including special biochemical examination of blood serum to determine the level of high-sensitivity C-reactive protein (CRP, mg/L) and lipid spectrum, including total cholesterol (GC, mmol/L), low-density lipoproteins (LDL, mmol/L), high-density lipoproteins (HDL, mmol/L), triglycerides (TG, mmol/L); urinalysis and instrumental examinations: electrocardiography (ECG), echocardiography (Echo-CG), R-graphy of chest organs, selective coronary angiography In addition to standard research methods, all patients will be determined molecular genetic parameters. Standard methods of investigation will be repeated after one year (2 points).

Preparation of DNA preparations. DNA extraction from blood was performed by phenol-chloroform extraction. Five to six volumes of buffer A (10 mM Tris-HCl, pH=7.5; 10 mM NaCl; 3 mM MgCl2) were added to 1 volume of blood sample and clots were rubbed in a homogenizer. After centrifugation at 2500g for 15 min, the precipitates were washed three times with buffer A and resuspended in 1 ml of buffer B (10 mM EDTA; 100 mM NaCl; 50 mM Tris-HCl, pH=8.5). After adding SDS to 0.5% and proteinase E to 200 μg/mL, the mixture was incubated for 12 hours at 56°C. Deproteinization was performed sequentially with phenol-chloroform mixture (1:1), water-saturated phenol, phenol-chloroform mixture (1:1), and chloroform. DNA was precipitated by adding NaCl solution to 1 M and 1 V isopropyl alcohol. After that, the solution was cooled for 1 h at -20 °C. The precipitate obtained by centrifugation on an Eppendorf microcentrifuge at 12000g for 15 min was washed three times with 75% ethanol followed by centrifugation for 5 min. 12000g and, after drying at 56 °C, dissolved in deinanilized water to a DNA concentration of 0.5 µg/μl.Genotyping of polymorphisms was performed using real-time PCR according to the manufacturer's protocol (TaqMan probes, Thermo Fisher Scientific, USA) on a StepOnePlus instrument. They were selected according to the results of international full genome-wide association studies (GWAS), which confirmed the association of these SNPs with coronary heart disease (CHD), an inflammatory process that plays a significant role in the progression of atherosclerosis.

Methods of statistical analysis. SPSS 22.0 software package will be used for statistical analysis of molecular-genetic data. The first stage will be to determine the frequencies of genotypes and alleles of the studied SNPs in the group of myocardial infarction patients with elevated values of cardiospecific markers and the comparison group, where cardiospecific markers will be within normal limits; then we will assess compliance of genotype frequencies with Hardy-Weinberg equilibrium in the control group (using the chi-square criterion). There will be a comparison of the levels of indicators such as age; cre-atinine level; diagnostic level of biomarkers of myocardial necrosis: MB creatine kinase and troponin, fatty acid binding protein (FABP); body mass index; waist circumference; serum C-peptide concentration; glycemia levels at admission and discharge; blood hemoglobin levels at admission and discharge; Systolic and diastolic blood pressure at admission; heart rate at admission; left ventricular ejection fraction value by echocardiography; serum HCMP concentration; lipidogram: serum concentration of low-density lipoproteins (LDL), high-density lipoproteins (HDL), total cholesterol, triglycerides; height, weight, body mass index, in carriers of different genotypes were performed after checking normality of distribution of these features by Kolmogorov-Smirnov test. If the traits would meet the criteria of normal distribution, a single-factor analysis of variance would be used. Significance of differences between two genotypic classes will be additionally checked using t-test for two independent samples. If a trait under study does not meet the criteria of normal distribution, comparison of the level of this trait in carriers of different genotypes will be performed using the Kruskal-Wallis test; the reliability of differences between the two genotypic classes will be additionally checked using the Mann-Whitney test for two independent samples. The association of SNPs with risk factors related to categorical variables will be tested with conjugation tables using Pearson chi-square test. In the case of four-field tables, comparison of samples by genotype and allele frequencies will use Fisher's exact two-sided criterion. The relative risk (OR - odds ratio) of disease outcome/risk factor presence for a particular allele or genotype will be calculated as odds ratio.

Influence of clinical, demographic, functional, metabolic, inflammatory parameters and myocardial necrosis markers on long-term prognosis will be assessed by odds ratio (0.95 confidence interval).

ELIGIBILITY:
Inclusion Criteria:

* who had had a type 1 myocardial infarction (MI) within two years prior to the study or had been diagnosed with CAD by selective coronary angiography: the presence of lumen stenosis of at least two coronary arteries of 50% or more and two (or more) additional cardiovascular events of the following: MI or unstable angina, emergency artery stenting, stroke, peripheral artery thrombosis, critical ischemia and lower limb amputation
* signed informed consent

Exclusion Criteria:

* patients with obstructive, dilated and restrictive cardiomyopathy, valve heart disease, malignant neoplasms, with acute inflammatory processes of the liver, kidneys, endocrine glands and other organs and systems, and chronic diseases in the phase of acute and incomplete remission; with diabetes mellitus type 1 and 2; atrial fibrillation of any type, severe hepatic and renal failure; chronic alcoholism and mental disorders, lack of signed voluntary informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort study included 202 patients with coronary heart disease. Group 1 included patients who had had myocardial infarction or unstable angina, emergency arterial stenting, stroke, peripheral artery thrombosis, critical ischemia, and lower extremity amputation within 2 years before study inclusion. Patients in the comparison group did not have these events. The influence of each of the studied parameters on the probability of fast progressing atherosclerosis was determined by factor and correlation analysis.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
death, MI, stroke | 2 years
  The analysis will be performed using the SPSS REGRESSION module

SECONDARY OUTCOMES:
total mortality | 1 year
  Statistical analysis of the prospective part of the study: the 2 study groups will be compared by endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Olga M. Parkhomenko, Study Chair — Novosibirsk State Medical University, Novosibirsk, Krasny pr 52, Russia
Locations (1):
- Novosibirsk State Medical University, Novosibirsk, Novosibirskaja Oblast' (oblast'), Russia

IPD SHARING:
Plan to Share IPD: No
gender, age, endpoints